CLINICAL TRIAL: NCT05960214
Title: Management of Patients With Thalassemia Minor and Breast Cancer at CardioOncology Outpatient Clinics: Age Quod Agis (AQUA)
Brief Title: Cardiac Management of Patients With Thalassemia Minor and Breast Cancer
Acronym: AQUA
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cafer Zorkun, Associate Professor, Istanbul University
Other Study IDs: COEXIST-3
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Thalassemia Minor; Heart Diseases
Keywords: Cardiotoxicity; Cancer treatment related cardiac dysfunctions
MeSH Terms: conditions — Breast Neoplasms; beta-Thalassemia; Heart Diseases; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 13 pts with BC+TM: Patients diagnosed with breast cancer and thalassemia minor
- 13 pts with BC: Patients diagnosed with breast cancer for comparison.

SUMMARY:
This retrospective study aimed to evaluate the demographic characteristics, clinical conditions in term of physical examination findings), functional status, and laboratory results of patients with thalassemia minor (TM) and breast cancer (BC) in order to identify any differences between the group with BC only.

Available data as anticancer treatment, comorbidities, weight and height will be combined to report body mass index (BMI) in kg/m2, systolic and diastolic blood pressure, heart rate, ECG, transthoracic echocardiography, blood count, lipid panels, glucose, kidney function tests, (N terminal) NT-proBNP, troponins, handgrip assessments, functional status were extracted from patients files and hospital electronic archives.

DETAILED DESCRIPTION:
Following data was extracted from files and hospital electronic records, and will be evaluated (at baseline, 3, 6, 9 and 12 months):

1. Physical examination findings (as pretibial edema, jugular venous distension, lung rales),
2. Clinically significant changes in cardiac function as determined by Left Ventricular Ejection Fraction (LVEF) measurements using transthoracic echocardiography,
3. Any changes in (N terminal) NT-ProBNP and troponin,
4. Any changes in manual handgrip measurements for both hands using hydraulic hand dynamometer,
5. Applied medications,

were extracted and will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of breast cancer, and thalassemia minor,
2. >18 years old,
3. Referred by oncologist for cardiac evaluation.
4. Patients with available cardiac evaluations data at baseline and during breast cancer treatment

Exclusion Criteria:

1. Patients without diagnosis of breast cancer, and thalassemia minor,
2. <18 years old,
3. Patients without any cardiac evaluations at baseline, and during cancer treatment.
4. Patients with history of any cardiotoxic treatment prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer and thalassemia minor and patients with breast cancer only.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of any rise in troponin | From enrollment to 12 months
  Troponin results from baseline and at 3, 6 and 12 months of cancer treatment .
Incidence of any rise in NT-ProBNP | From enrollment to 12 months
  NT-ProBNP results from baseline and at 3, 6 and 12 months of cancer treatment .
Incidence of any reduction in LV | From enrollment to 12 months
  Echocardiographic measurements of Left ventricle (LV) ejection fraction from baseline and at 3, 6 and 12 months of cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Cafer Zorkun, MD PhD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data underlying this article cannot be shared due to privacy concerns for the individuals who participated in the study. However, after obtaining proper permission from the IRB (Institutional Review Board), a summary of the data at the aggregate level, without individual identifiers, will be made available.